CLINICAL TRIAL: NCT06894914
Title: Moving More: Supporting Uptake of Evidence for Physical Activity in Older Adults With Complex Health Care Needs
Brief Title: Supporting Uptake of Evidence for Physical Activity in Older Adults With Complex Health Care Needs
Acronym: Moving_More
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Arthritis Research Centre of Canada (Other)
Responsible Party: Principal Investigator, Linda Li, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: H24-03597
Record Dates: First submitted 2025-02-23; First posted 2025-03-25 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Frailty
Keywords: Physiotherapy; Physical activity; Sleep; Counselling
MeSH Terms: conditions — Frailty; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 24-hour Activity Counselling (Experimental): Participating physiotherapists will be trained to deliver counselling that focuses on increasing moderate-to-vigorous physical activity, with a balance of activity, rest and sleep in a 24-hour day.
  Patients (n=4) of these physiotherapists will receive the 24-hour Activitiy Counselling
  Interventions: Behavioral: 24-hour Activity Counselling
- Current Physical Activity Counselling (Active Comparator): Participating physiotherapists will continue delivering counselling that focuses on achieving 150 minutes/week of moderate-to-vigorous physical activity, which is the current practice.
  Patients (n=4) of these physiotherapists will receive the Current Physical Activitiy Counselling
  Interventions: Behavioral: 24-hour Activity Counselling

INTERVENTIONS:
Behavioral: 24-hour Activity Counselling — Physiotherapists will participate in the self-paced brief action planning (BAP) online training (2-4 hours long), followed by 2-3 hours of practice and feedback over the phone with an experienced BAP instructor. In addition, they will attend a 2-hour session with the research team on training around on prescribing physical activity while balancing with rest and sleep.
  Once training is complete the PT can start implementing the counselling approach with the older adult patients.

SUMMARY:
Physically frail older adults often have chronic conditions that contribute to a higher chance of them being limited in daily activities and becoming dependent. Physical activity can help to better manage chronic conditions and prevent frailty. In this project, the counselling approach using the new Canadian 24-hour Movement Guidelines will be adapted for older adults at an early state of frailty. This new approach will be tested against the one in current use by physiotherapists. This ethics application will address the pilot implementation evaluation, including interviews and focus groups, conducted to refine the new approach.

DETAILED DESCRIPTION:
Rationale:

Physical activity is effective in preventing the progression of frailty and further disability in community-dwelling frail older adults. It is also effective in mitigating the progression of chronic conditions associated with physical frailty. Despite the benefits, many older adults in the early state of frailty and with chronic conditions are not sufficiently active. Current delivery of physical activity recommendations can be improved by applying the new Canadian 24-hour Movement Guidelines. These guidelines promote a balance of activity, rest and sleep as they play an important role for better overall health and quality of life regardless of health conditions. With advanced training in complex chronic conditions and physical activity promotion, physiotherapists (PTs) are well-suited to adapt and integrate activity counselling, based on the 24-hour Movement Guidelines, in their clinical practice.

Aim:

to assess implementation context, feasibility, and preliminary effect of the 24-hour Approach against a current goal-oriented counselling approach (i.e., focus on achieving 150 minutes/week of MVPA).

Previous Work:

A PT-led goal-oriented counselling program was previously evaluated for older adults with osteoarthritis. In 2 randomized controlled trials (RCTs), compared to controls, this program was shown to improve time spent in Moderate/Vigorous Physical Activity (MVPA) in participants after 8 weeks (n=61; 25.6 mins/day; 95% CI. 9) and 13 weeks (n=51; 13.1 mins/day; 95% CI. 5). This current approach has been modified for remote delivery during the COVID-19 pandemic.

Research Design & Data Analysis:

This is a multi-method study. PTs and their patients across Canada who have participated in the co-development of the 24-hour Approach will be invited to participate. The 24-hour Approach will be assessed in a randomized pilot study with 20 PTs and their patients (each PT will treat 4 older adult patients) who will be assigned to one of the groups:

1. Current Approach (focus on achieving 150 min/week of MVPA).
2. 24-hour Approach (focus on increasing MVPA with a balance of activity, rest and sleep in a day).

Guided by the RE-AIM framework, Reach will be assessed by comparing characteristics of older adult participants with those who are eligible yet decline to participate. Effect (Preliminary) will be evaluated at the older adult level. Adoption will be assessed by comparing the demographic and practice characteristics between the participating PTs and those who are eligible but have not enrolled. Implementation will be assessed by PT interviews when they complete their sessions with all 4 older adult patients. To assess Maintenance, PTs will be interviewed at 12 months about if/how they continue using their assigned counselling strategy after the study. Results will inform a full RCT and future scale-up.

Significance:

Results will provide necessary knowledge to inform how to improve uptake of physical activity recommendations in ways that are sensitive to the health needs of older adults and their life context.

ELIGIBILITY:
Physiotherapists:

Inclusion Criteria:

* Eligible PTs are those who self-report at least 40% of their caseload is working with older adults and practice in the in the Greater Vancouver Area. In addition, they are willing to:

  1. participate in online training for the assigned physical activity counselling strategy
  2. be randomised to one of the counselling groups.

Exclusion Criteria:

* Those who do not meet the Inclusion Criteria

Older adults:

Inclusion Criteria:

1. are age > 65 years
2. live in the community
3. have 1 or 2 of the deficits in the CHS index
4. have > 1 chronic conditions
5. are able to walk 3 metres with or without an assistive device
6. have a Mini-Mental State Examination score > 24/30
7. do not have a diagnosed psychiatric condition (e.g., depression)
8. understand, speak and read English proficiently
9. are willing to have their physiotherapy sessions audio-recorded
10. are able to provide written informed consent.

Exclusion Criteria:

* Those who do not meet the Inclusion Criteria

Max Age: 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Patient's daily time in moderate/vigorous physical activity (minutes/day) | 6 months
  Minutes spent in moderate/vigorous physical activity per day

SECONDARY OUTCOMES:
Patient's daily time in moderate/vigorous physical activity (minutes/day) | 12 months
  Minutes spent in moderate/vigorous physical activity per day
Patient's daily time in light physical activity (minutes/day) | 6 months
  Minutes spent in light physical activity per day
Patient's daily time in light physical activity (minutes/day) | 12 months
  Minutes spent in light physical activity per day
Patient's daily time in sedentary behaviour (minutes/day) | 6 months
  Minutes spent in sedentary behaviour per day
Patient's daily time in sedentary behaviour (minutes/day) | 12 months
  Minutes spent in sedentary behaviour per day
Patient's daily time sleeping (minutes/day) | 6 months
  Minutes spent sleeping per day
Patient's daily time sleeping (minutes/day) | 12 months
  Minutes spent sleeping per day
The score of cardiovascular Health Study (CHS) index (Patient outcome) | 6 months
  multidimensional measure of physical frailty (0-5 points; lower = better)
  1. Weight Loss: Lost > 10 pounds unintentionally in last year
  2. Exhaustion Self-report of either of:
     i. felt that everything I did was an effort in the last week ii. could not get going in the last week
  3. Weakness Grip strength: Lowest 20% adjusted for sex and body mass index
  4. Low Physical Activity Women: Kcal < 270 on activity scale (18 items)§ Men: Kcal < 383 on activity scale (18 items)§
  5. Slowness Walking time: Slowest 20% adjusted by sex and height
  "Yes" to each of the above is 1 point.
The Cardiovascular Health Study (CHS) index score (Patient outcome) | 12 months
  multidimensional measure of physical frailty (0-5 points; lower = better)
  1. Weight Loss: Lost > 10 pounds unintentionally in last year
  2. Exhaustion Self-report of either of:
     i. felt that everything I did was an effort in the last week ii. could not get going in the last week
  3. Weakness Grip strength: Lowest 20% adjusted for sex and body mass index
  4. Low Physical Activity Women: Kcal < 270 on activity scale (18 items)§ Men: Kcal < 383 on activity scale (18 items)§
  5. Slowness Walking time: Slowest 20% adjusted by sex and height
  "Yes" to each of the above is 1 point.
Short Physical Performance Battery (SPPB; 0-12; higher = better; Patient outcome) | 6 months
  Short Physical Performance Battery (SPPB) is a standardized measure of lower extremity physical performance that includes walking, balance, and strength tasks, and has been used in a broad range of RCTs and epidemiological studies of aging. A low SPPB score is a strong risk factor for institutionalization, morbidity, mortality, and disability in initially non-disabled older persons. Participants are assessed on performances of standing balance, 4-m walking, and sit-to-stand. Each component is rated out of 4 points, for a maximum of 12 points.
Short Physical Performance Battery (SPPB; 0-12; higher = better; Patient outcome) | 12 months
  Short Physical Performance Battery (SPPB) is a standardized measure of lower extremity physical performance that includes walking, balance, and strength tasks, and has been used in a broad range of RCTs and epidemiological studies of aging. A low SPPB score is a strong risk factor for institutionalization, morbidity, mortality, and disability in initially non-disabled older persons. Participants are assessed on performances of standing balance, 4-m walking, and sit-to-stand. Each component is rated out of 4 points, for a maximum of 12 points.
Gait speed (meters/second; Patient outcome) | 6 months
  Gait speed will be calculated by dividing the 4-meter walk with the time to complete the walk
Gait speed (meters/second; Patient outcome) | 12 months
  Gait speed will be calculated by dividing the 4-meter walk with the time to complete the walk
Grip strength (in kg) of the dominant hand (Patient outcome) | 6 months
  Grip strength (in kg) of the dominant hand will be measured using a digital Jamar isometric hand dynamometer; three measures will be acquired and averaged.
Grip strength (in kg) of the dominant hand (Patient outcome) | 12 months
  Grip strength (in kg) of the dominant hand will be measured using a digital Jamar isometric hand dynamometer; three measures will be acquired and averaged.
EuroQol-5D-5 Level version (EQ-5D-5L; Patient outcome) | 6 months
  measure Health-Related Quality of Life. EQ-5D-5L is a generic preference-based utility measure composed of 5 domains of health (mobility, self-care, usual activities, pain, and anxiety/depression). Each domain contains 5 levels ('1' indicating no problem; '5' indicating major problem).
EuroQol-5D-5 Level version (EQ-5D-5L; Patient outcome) | 12 months
  measure Health-Related Quality of Life. EQ-5D-5L is a generic preference-based utility measure composed of 5 domains of health (mobility, self-care, usual activities, pain, and anxiety/depression). Each domain contains 5 levels ('1' indicating no problem; '5' indicating major problem).
Self-Reported Habit Index (Patient outcome) | 6 months
  A multi-item measure rated on a 7-point Likert scale that evaluates characteristics of habitual behavior
Self-Reported Habit Index (Patient outcome) | 12 months
  A multi-item measure rated on a 7-point Likert scale that evaluates characteristics of habitual behavior

CONTACTS AND LOCATIONS:
Overall Officials: Linda Li, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Arthritis Research Canada, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to share individual participant data from this clinical trial, including demographics, baseline characteristics, primary outcome measures, and key secondary outcomes, with qualified researchers upon request after the study results have been published.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: TBA
Access Criteria: Data will be provided in a de-identified format through a secure online repository, and access will require submission of a research proposal outlining the intended analysis and relevant ethics approvals.